CLINICAL TRIAL: NCT02982330
Title: Impact of a Low Carbohydrate Breakfast on Glucose Control in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Dr Jonathan P Little, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H16--00377
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Carbohydrate Breakfast (Experimental): Breakfast composition containing <10% carbohydrate, 75% fat, 15% protein Matched calories
  Interventions: Behavioral: Low Carbohydrate Breakfast; Behavioral: Guidelines Breakfast
- Guidelines Breakfast (Active Comparator): Breakfast composition containing 55% carbohydrate, 30% fat, 15% protein Matched calories
  Interventions: Behavioral: Low Carbohydrate Breakfast; Behavioral: Guidelines Breakfast

INTERVENTIONS:
Behavioral: Low Carbohydrate Breakfast — A low carbohydrate breakfast containing <10% carbohydrate, ~75% fat, and 15% protein. Matched for calories to the active comparator arm.
Behavioral: Guidelines Breakfast — A low fat breakfast containing ~55% carbohydrate, <30% fat, and 15% protein. Matched for calories to the experimental arm.
  Other Names: Low-fat Breakfast

SUMMARY:
Large glucose excursions at breakfast are prevalent in type 2 diabetes and can contribute to sustained hyperglycaemia across the day. Lowering consumption of dietary carbohydrate is known to reduce post-meal glucose excursions but it is unknown whether lowering the carbohydrate at breakfast only will impact subsequent post meal glucose excursions throughout the day. The aim of this study is to examine, under free living conditions and using typical dietary patterns, whether eating a breakfast low in carbohydrate can lower daily post-meal glycemia when compared to consuming a low-fat breakfast (per the current diabetes guidelines).

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed Type 2 Diabetes (>6 months)

Exclusion Criteria:

* Exogenous Insulin
* A1c > 9%
* Cardiovascular, liver, or renal other disease
* Breakfast and meal skippers

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-11; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Incremental area under the glucose curve (continuous glucose monitor) | 24 hour (one day)

SECONDARY OUTCOMES:
Mean Blod Glucose (continuous glucose monitor) | 24 hours (one day)

OTHER OUTCOMES:
Glycemic Variability (continuous glucose monitor) | 24 hours (one day)
Satiety VAS 100 | Before and after meals (one day)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Little, PhD, Principal Investigator — UBC Okanagan
Locations (1):
- University of British Columbia, Okanagan., Kelowna, British Columbia, Canada

REFERENCES:
- [Derived] Chang CR, Francois ME, Little JP. Restricting carbohydrates at breakfast is sufficient to reduce 24-hour exposure to postprandial hyperglycemia and improve glycemic variability. Am J Clin Nutr. 2019 May 1;109(5):1302-1309. doi: 10.1093/ajcn/nqy261. PMID 30968140